CLINICAL TRIAL: NCT01774877
Title: Efficacy and Safety of Xinfeng Capsule in the Treatment of Rheumatoid Arthritis (RA):A Randomized, Double-blind, Double-dummy, Multi-center Trial
Brief Title: A Clinical Study of Xin'an Medicine in the Treatment of Bi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Jian, professor，Chief Physician, The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012BAI26B02
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Rheumatoid Arthritis
Keywords: xinfeng capsule;; rheumatoid arthritis (RA);; randomized;; double-blind;
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — xinfeng; Leflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xinfeng capsule & placebo (Experimental): 1. Xinfeng capsule:Three each time, 3 times a day, Oral,for 3 months
  2. placebo(for leflunomide): 10 mg each time, 1 time a day, Oral,for3 months
  Interventions: Drug: Xinfeng capsule
- leflunomide & placebo (Active Comparator): 1. leflunomide :10mg each time, one time a day, by mouth,for 3 months
  2. placebo(for xinfeng capsule):Three each time, 3 times a day, Oral,for3 months
  Interventions: Drug: leflunomide

INTERVENTIONS:
Drug: Xinfeng capsule — Xinfeng capsule:Three each time, 3 times a day, Oral,for 3 months; placebo(for leflunomide):10mg each time, 1 time a day, Oral,for 3 months; Participants will continue on the stable dose of glucocorticoids and NSAIDs that they were receiving prior to study entry
  Arms: Xinfeng capsule & placebo
Drug: leflunomide — leflunomide :10mg each time, one time a day, Oral,for 3 months; placebo(for xinfeng capsule):Three each time, 3 times a day, Oral,for 3 months; Participants will continue on the stable dose of glucocorticoids and NSAIDs that they were receiving prior to study entry
  Arms: leflunomide & placebo

SUMMARY:
Bi Syndrome is one of Traditional Chinese Medicine（TCM）name, It means an obstruction in Chinese,and it refers the syndrome characterized by the obstruction of qi and blood in the meridians due to the invasion of external pathogenic wind,cold and dampness, manifested as soreness, pain, numb,etc. Bi Syndrome contains Rheumatoid arthritis(RA). RA is a chronic disease affecting more than 20 million people in the world.It is one of the most common forms of autoimmune disease. Xin'an Medicine is one of Traditional Chinese Medicine which originated from AnHui. Xinfeng Capsule developed according to the Xin'an medicine theory ,and it has long been adopted for treatment of rheumatoid arthritis (RA). The study is aimed to evaluate the effectiveness and safety of Xinfeng Capsule in the treatment of RA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA, classified by American Rheumatism Association 1987 revised criteria.
* According with the Zheng diagnosis of Traditional Chinese Medicine.
* age from 18 to 65 years.
* For patients currently receiving non-steroidal anti-inflammatory drugs (NSAIDs): Treatment at a stable dose during last 4 weeks prior to screening，or Patients do not take NSAIDs at least 1 weeks prior to screening.
* Patients not taking DMARDs at least 4 weeks prior to screening.
* Patients taking corticosteroids (≤15mg prednisone or Equivalent) ≥4 weeks before entering the trial.
* Patients agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients have received intra-articular or systemic corticosteroid injection within 4 weeks of screening.
* Patients have high disease activity (DAS28-3 scores> 5.1).
* Patients have diagnosed any other chronic inflammatory disease or connective tissue disease like sicca syndrome（SS）, systemic lupus erythematosus (SLE)etc;
* Patients with sever diseases in Cardiovascular, brain, lung, liver, kidney and hematopoietic system ;
* Patients who are pregnant or nursing mothers or Psychiatric patients.
* Patients with active gastroduodenal ulcer or gastritis which caused by long-term use of NSAIDs;
* The patient who has known hypersensitivity to trial medicine .
* Patients have participated in other clinical trials within 4 weeks of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
ACR20 (American College of Rheumatology (ACR) criteria of 20% improvement in symptoms ) | baseline,week4,week8,week12
  ACR20 used for evaluating the efficacy of rheumatoid arthritis (RA).

SECONDARY OUTCOMES:
ACR50 (American College of Rheumatology (ACR) criteria of 50% improvement in symptoms ) | baseline,week4,week8，week12
  ACR50 used for evaluating the efficacy of rheumatoid arthritis (RA).
ACR70 (American College of Rheumatology (ACR) criteria of 70% improvement in symptoms ) | baseline,week4,week8，week12
  ACR50 used for evaluating the efficacy of rheumatoid arthritis (RA).
Patterns based on Chinese medicine(CM)symptoms | baseline,week4,week8，week12
Disease Activity Scale (DAS)28 | baseline,week4,week8, week12
Rheumatoid arthritis (RA) biomarkers | baseline, week12
  Rheumatoid arthritis (RA) biomarkers,including rheumatoid factor (RF), erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) ,anti-cyclic citrullinated peptide (anti-CCP) antibodies, IgG、IgA、IgM, d-dimer, the coagulation function tests
Life Quality Assessment | baseline,week12
  Life Quality Assessment,including Health Assessment Questionnaire (HAQ), Self-rating depression scale(SDS), Self-rating anxiety scale(SAS),quality of life Questionnaire with rheumatoid arthritis.
x-rays of the hands and wrists | baseline,week12

CONTACTS AND LOCATIONS:
Overall Officials: liu jiu, doctor, Principal Investigator — The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Locations (3):
- China (3):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - The first affiliated hospital of anhui medical university, Hefei, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui

REFERENCES:
- [Derived] Liu J, Wang Y, Huang C, Xu J, Li Z, Xu L, He L, Sun Y, Wang Y, Xu S, Zhao P, Mao T, Tan B, Zhu F, Zhang P, Fang L. Efficacy and safety of Xinfeng capsule in patients with rheumatoid arthritis: a multi-center parallel-group double-blind randomized controlled trial. J Tradit Chin Med. 2015 Oct;35(5):487-98. doi: 10.1016/s0254-6272(15)30130-8. PMID 26591677
- [Derived] Liu J, Huang CB, Wang Y, Xu GQ, Cheng YY, Feng YX, Liu L, Qi YJ. Chinese herbal medicine Xinfeng Capsule in treatment of rheumatoid arthritis: study protocol of a multicenter randomized controlled trial. J Integr Med. 2013 Nov;11(6):428-34. doi: 10.3736/jintegrmed2013059. PMID 24299607